CLINICAL TRIAL: NCT03824964
Title: An Observational Clinical Study on the Safety and Efficacy of Anti-CD19/CD22 CAR NK Cells in Relapsed and Refractory B Cell Lymphoma
Brief Title: Study of Anti-CD19/CD22 CAR NK Cells in Relapsed and Refractory B Cell Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19/CD22 CAR NK-BJZL-01
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Refractory B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Anti-CD19/CD22 CAR NK Cells — Total dose of 50-600 thousand /kg Anti-CD19/CD22 CAR NK cells will be administered at day0

SUMMARY:
This is a single-centre, single-arm and open-label study to investigate the safety and efficacy of anti CD19/CD22 CAR NK cells in patients with relapsed refractory B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. CD19(+) CD22(+) B cell lymphoma confirmed by pathological immunohistochemistry or flow cytometry
2. Previously accepted ≥ first-line regimen chemotherapy
3. Unconditional acceptance of hematopoietic stem cell transplantation or recurrence after hematopoietic stem cell transplantation
4. Over 18 years old and under 70 years old
5. The expected survival period is more than 3 months.
6. ECOG≤2
7. Important organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥50%, no abnormal electrocardiogram; blood oxygen saturation ≥90%; creatinine clearance ≥40 mL/min; ALT and AST≤3 times normal range, Total bilirubin ≤ 2.0 mg / dL;
8. Blood routine: Hgb≥80 g/L, ANC≥1×109/L, PLT≥50×109/L;
9. The pregnancy test for women of childbearing age must be negative; both men and women must agree to use effective contraception during the treatment period and for the following 1 year.
10. Measurable target lesion

Exclusion Criteria:

1. Patients with extramedullary relapse
2. Burkitt's lymphoma/leukemia
3. Previously received gene product treatment, anti-CD19/anti-CD3 treatment, or any anti-CD19/CD22 treatment;
4. Liver and kidney function:

   * Total bilirubin > 2 x ULN (Gilbert Syndrome > 3 x ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 3 × ULN
   * Serum creatinine clearance >60 mL/min
5. Serological examination:

   * Absolute neutrophil count (ANC) <0.75x109/L
   * Platelet count (PLT) <50x109/L
6. Active hepatitis B (HBV-DNA > 1000 copies / mL), hepatitis C, or uncontrolled infection
7. GVHD ≥ 2 or anti-GVHD treatment
8. IM19 CAR NK cells received allogeneic cell therapy within 6 weeks before infusion, such as donor lymphocyte infusion;
9. Subject received the most recent treatment (release, chemotherapy, or other) less than 4 weeks
10. Active CNS disease (tumor cells in CSF, but < 5 WBCs/mL can be included);
11. Intracranial hypertension or unconsciousness; respiratory failure; diffuse vascular internal coagulation
12. Creatinine > 1.5 times normal upper limit or ALT / AST > 3 times normal upper limit or bilirubin > 2 times normal upper limit
13. New York Heart Association (NYHA) graded above or above
14. Uncontrollable diabetes
15. Suffering from other uncontrolled diseases, the researchers believe that it is not suitable for joining
16. Any situation that the investigator believes may increase the risk of the subject or interfere with the test results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.0 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment.